CLINICAL TRIAL: NCT00644930
Title: The Efficacy of Non-Invasive Positive Pressure Ventilation in ARDS: A Controlled Cohort Study
Brief Title: Non-Invasive Positive Pressure Ventilation and Adult Respiratory Distress Syndrome (ARDS)
Acronym: NPPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Dr. Irfan Ucgun, Eskisehir Osmangazi University, Department of Chest Diseases
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISRCTN73824458; ISRCTN73824458
Record Dates: First submitted 2008-03-14; First posted 2008-03-27 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2008-03

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS,; noninvasive ventilation,; intubation,; mortality,; intensive care
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): ARDS patients in the NPPV group showing no indications for urgent intubation received NPPV in addition to standard medical therapy, and those with indications were intubated.
  Interventions: Device: the application of NPPV
- 2 (Active Comparator): Patients in the standard therapy group without indications for urgent intubation were only given standard medical therapy (such as oxygen, antibiotics, and bronchodilators), and IMV through an endotracheal tube was applied when intubation criteria were met.
  Interventions: Device: invasive ventilation

INTERVENTIONS:
Device: the application of NPPV — ARDS patients in the NPPV group showing no indications for urgent intubation received NPPV in addition to standard medical therapy, and those with indications were intubated. BIPAP Vision machine (Respironics, PA, USA) were used for NPPV.
  Other Names: NPPV group
  Arms: 1
Device: invasive ventilation — Standard therapy group (invasive ventilation). Patients in need of endotracheal intubation were mechanically ventilated with Amadeus (Hamilton, Via Nova, Switzerland) and Esprit (Respironics, PA, USA) ventilators in the assist-control or synchronized intermittent mandatory ventilation (SIMV) mode.
  Other Names: Standard therapy group
  Arms: 2

SUMMARY:
Background and objective: To determine the efficacy of non-invasive positive pressure ventilation (NPPV) and its effects upon intubation rate and mortality in ARDS.

DETAILED DESCRIPTION:
Methods: This study was performed in the respiratory intensive care unit (ICU) at a university hospital. 20 patients who achieved the diagnostic criteria for ARDS were included. The patients were prospectively allocated into two groups: a standard therapy group and a NPPV group. Invasive mechanical ventilation indications had been determined before the study. Invasive ventilation was applied to those who in need of intubation, while those given intubation received a standard medical treatment.

ELIGIBILITY:
Inclusion Criteria:The following criteria indicated immediate intubation was needed:

1. Apne or respiratory pauses with loss of consciousness or gasping for breath or imminent respiratory arrest.
2. Inability to increase the patient's PaO2 to more than 40 mmHg and SpO2 to more than 80% with a FiO2>0.6.
3. Inability to increase the patient's pH levels above 7.35, and development of blurred consciousness and confusion (Glasgow Coma Scale <9) due to respiratory acidosis despite all the support given.
4. Instability of the patient's hemodynamic parameters (such as systolic blood pressure <80 mmHg or heart rate <50 beats/minute lasting >1 hour despite fluid resuscitation).

Exclusion Criteria:Contraindications for NPPV include:

1. The need for urgent intubation.
2. The need for frequent aspiration due to excessive secretions (more frequent than 15 min.).
3. Inability of the patient to adapt himself / herself to the device or unwillingness to undergo NPPV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-08; Primary Completion 2005-09 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Intubation rate | 48 hours

SECONDARY OUTCOMES:
Hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Irfan Ucgun, Ass Prof Dr, Study Chair — Eskisehir Osmangazi University, Medical Faculty, Department of Chest Dis.
Locations (1):
- Eskisehir Osmangazi University, Medical Faculty,, Eskişehir, Merkez, Turkey (Türkiye)

REFERENCES:
- [Result] Rana S, Jenad H, Gay PC, Buck CF, Hubmayr RD, Gajic O. Failure of non-invasive ventilation in patients with acute lung injury: observational cohort study. Crit Care. 2006;10(3):R79. doi: 10.1186/cc4923. Epub 2006 May 12. PMID 16696863
- [Result] Liesching T, Kwok H, Hill NS. Acute applications of noninvasive positive pressure ventilation. Chest. 2003 Aug;124(2):699-713. doi: 10.1378/chest.124.2.699. PMID 12907562
- [Result] Antonelli M, Conti G, Esquinas A, Montini L, Maggiore SM, Bello G, Rocco M, Maviglia R, Pennisi MA, Gonzalez-Diaz G, Meduri GU. A multiple-center survey on the use in clinical practice of noninvasive ventilation as a first-line intervention for acute respiratory distress syndrome. Crit Care Med. 2007 Jan;35(1):18-25. doi: 10.1097/01.CCM.0000251821.44259.F3. PMID 17133177